CLINICAL TRIAL: NCT05054985
Title: Guo's Renovisceral Artery Reconstruction-1: a Prospective, Multicenter, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of a Multi-branched Stent Graft System for Thoracoabdominal Aortic Aneurysm (GUARANTEE Study)
Brief Title: Safety and Efficacy of a Multi-branched Thoracoabdominal Stent Graft System for Thoracoabdominal Aortic Aneurysm.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ-TAAA-01
Record Dates: First submitted 2021-09-07; First posted 2021-09-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Thoracoabdominal Aortic Aneurysms
Keywords: Guo's Visceral Arteries Reconstruction; Multi-branched Thoracoabdominal Stent Graft System; Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Patients with thoracoabdominal aortic aneurysms, and passed the screening and signed the informed consent form.
  Interventions: Device: Multi-Branched Thoracoabdominal Stent Graft System

INTERVENTIONS:
Device: Multi-Branched Thoracoabdominal Stent Graft System — Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with multi-branched thoracoabdominal stent graft system .

SUMMARY:
Evaluation of the safety and efficacy of a multi-branched thoracoabdominal stent graft system for thoracoabdominal aortic aneurysm.

DETAILED DESCRIPTION:
The study is mainly for patients with thoracoabdominal aortic aneurysms, and all subjects who signed the informed consent and passed the screening will be enrolled. Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with multi-branched thoracoabdominal stent graft system. Patients will be followed up at discharge, 1 month, 6 months, 12 months after the implantation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 80 years old;
2. Diagnosed as thoracoabdominal aortic aneurysm (based on modified Crawford classification and 2019 European Guidelines for the Treatment of Aortic aneurysm) and should meet at least one of the following conditions;

   1. Maximum diameter of thoracoabdominal aortic aneurysm>50mm;
   2. The diameter has increased by more than 5mm in recent 6 months or the by more than 10mm in recent 1 year;
3. anatomical criteria

   1. The proximal anchoring region (aorta or implanted graft) was 17~36 mm in diameter and ≥25 mm in length;
   2. Distal anchoring region (aorta or implanted graft): If the distal anchoring region is in the iliac artery, the anchoring region has a diameter range of 7~25 mm and a length of ≥15 mm; If the distal anchoring area is in the abdominal aorta, the diameter of the anchoring area ranges from 12~36mm and the length≥ 20mm;
   3. The diameter of the vessel anchoring area of the visceral branch ranges from 6~13 mm and the length ≥15 mm;
   4. The diameter of renal artery anchoring area ranges from 4.5~9mm, and the length ≥15 mm;
   5. Appropriate iliac, femoral and upper limb artery access;
4. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent, and are willing to complete the follow-up according to the requirements of the protocol;

Exclusion Criteria:

1. Hemodynamically unstable patients with ruptured thoracoabdominal aortic aneurysms;
2. Thoracoabdominal aortic dissection;
3. Mycotic or infectious thoracoabdominal aortic aneurysm;
4. Patients whose systemic or local infection may increase the risk of intravascular graft infection;
5. Superior mesenteric, celiac, or renal artery occlusion;
6. Requiring simultaneous coverage and embolization of bilateral internal iliac arteries;
7. Severe stenosis, calcification, or mural thrombus in the anchoring area of the stent tend to have difficulty in attachment of the stent-graft or affect the patency of the stent;
8. A history of acute coronary syndrome within 6 months; Acute coronary syndrome is defined as an acute ischemic syndrome of the heart resulting from the rupture or erosion of unstable intracoronary atherosclerotic plaques followed by fresh thrombosis, including ST-segment elevation myocardial infarction, non-ST-segment elevation myocardial infarction, and unstable angina pectoris.
9. Transient ischemic attack (TIA) or ischemic/haemorrhagic stroke within 3 months;
10. Preoperative liver renal function abnormalities (ALT or AST ≥ 5 times the upper limit of normal value), or serum creatinine ≥ 150 μmol/L;
11. Severe pulmonary insufficiency who cannot tolerate general anaesthesia;
12. Severe coagulation dysfunction;
13. Undergone major surgical or interventionic surgery within 30 days before surgery;
14. A history of allergy to contrast agents, anticoagulants, antiplatelet drugs, stents, and conveyor materials (nitinol, polyester, PTFE, nylon);
15. Connective tissue diseases such as systemic lupus erythematosus, Marfan's syndrome, Adam's syndrome, or Behcet's disease;
16. takayasu arteritis;
17. Serious vital organ dysfunction or other serious disease;
18. Planning pregnancy, pregnancy, or breastfeeding;
19. Patients who participated in other clinical trials and was not discontinued or withdrawn within the first 3 months of the screening period of this trial.
20. Life expectancy less than 1 year;
21. Patients who, in the judgment of the investigator, are not eligible for endotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint: The incidence of Major Adverse events (MAE) within 30 days after procedure. | Within 30 days after procedure
  Major Adverse Event (MAE) was defined as all-cause death, liver failure, intestinal necrosis, kidney failure, stroke, permanent paraplegia, myocardial infarction, and respiratory failure.
Primary efficacy endpoint: Success rate of thoracoabdominal aortic aneurysm treatment 12 months after procedure. | 12 months after procedure.
  Successful treatment of thoracoabdominal aortic aneurysm is a composite index that needs to meet the following indicators at the same time: Immediate technical success (immediate technical success refers to the successful delivery system to a predetermined location, the successful deployment of the system and the safe withdrawal of the delivery system from the body and no type I/III endoleak), no secondary surgical intervention related to thoracoabdominal aortic aneurysms 12 months after procedure (due to aneurysm rupture, continuous enlargement, stent displacement, type I/III endoleak, branch stenosis/ Second surgery caused by occlusion) .

SECONDARY OUTCOMES:
aneurysmal enlargement at 6 and 12 months postoperatively | 6 and 12 months postoperatively
  aneurysmal enlargement defined as a maximum aortic diameter increase of > 5 mm relative to preoperative computed tomography angiography (CTA)
type I/III endoleak at 6 and 12 months postoperatively | 6 and 12 months postoperatively
stent graft migration at 6 and 12 months postoperatively | 6 and 12 months postoperatively
renovisceral artery patency rate at 6 and 12 months postoperatively | 6 and 12 months postoperatively
reintervention secondary to TAAA progression at 6 months, 12 months, and 2-5 years postoperatively. | 6 months, 12 months, and 2-5 years postoperatively.
delivery system-related complications during the procedure and within 30 days postoperatively, including conversion to open surgery, and any hemorrhage, hematoma, or pseudoaneurysm of the arterial access | during the procedure and within 30 days postoperatively
all-cause mortality at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
TAAA-related mortality at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
device-related adverse events at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively
severe adverse events resulting in death or serious deterioration of health at 6 months, 12 months, and 2-5 years postoperatively | 6 months, 12 months, and 2-5 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data will be shared for scientific purposes after the completion of the clinical trial. However, patients' electronic records and any CTA files are outside the scope of our data sharing policy. Researchers wanting to request data can submit a detailed application to the investigators. Data will be released depending on the scientific quality of the submitted request.

REFERENCES:
- [Derived] Ge Y, Zhang H, Rong D, Liu F, Jia X, Xiong J, Ma X, Wang L, Fan T, Guo W. Protocol for GUo's renovisceral Artery reconstruction-1: a prospective, multicentre, single-arm clinical trial to evaluate the safety and efficacy of a multibRANched sTEnt graft systEm for thoracoabdominal aortic aneurysm (GUARANTEE study). BMJ Open. 2022 Mar 23;12(3):e059401. doi: 10.1136/bmjopen-2021-059401. PMID 35321900